CLINICAL TRIAL: NCT06037122
Title: Efficacy and Safety Evaluation of Bismuth-containing Quadruple Therapies Based on Low-dose Vonoprazan in the Initial Treatment of Helicobacter Pylori Infection: a Retrospective Study
Brief Title: Efficacy of Low-dose Vonoprazan for Helicobacter Pylori Eradication
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-0674
Record Dates: First submitted 2023-09-07; First posted 2023-09-14 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-08

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter Pylori; quadruple regimen; vonoprazan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- group R-BID: rabeprazole 10mg, amoxicillin 1000 mg, clarithromycin 500 mg, bismuth pectin 200 mg or bismuth potassium citrate 220mg twice daily, all drugs given for 14 days
- group V-BID: vonoprazan 20mg, amoxicillin 1000 mg, clarithromycin 500 mg, bismuth pectin 200 mg or bismuth potassium citrate 220mg twice daily, all drugs given for 14 days
- group V-QD: vonoprazan 20mg once daily, amoxicillin 1000 mg, clarithromycin 500 mg, bismuth pectin 200 mg or bismuth potassium citrate 220mg twice daily, all drugs given for 14 days

SUMMARY:
The primary objective of this retrospective study was to assess the efficacy and safety of a bismuth quadruple regimen of a low-dose potassium-competitive acid blocker versus a standard-dose potassium-competitive acid blocker and a standard-dose proton pump inhibitor combined with amoxicillin and clarithromycin as the initial treatment of Helicobacter pylori infection.

DETAILED DESCRIPTION:
Helicobacter pylori (H. pylori) infection is closely associated with a variety of diseases including chronic gastritis, peptic ulcer, and gastric cancer. Adequate acid suppression is essential for H. pylori eradication therapy. Potassium-competitive acid blocker (P-CAB) vonoprazan (VPZ) has faster, stronger, and longer-lasting acid inhibition and plays an important role in H. pylori treatment. 2022 Chinese national clinical practice guideline on Helicobacter pylori eradication treatment recommended for the first time a quadruple regimen of bismuth containing P-CAB for H. pylori eradication, in which P-CAB was administered as VPZ 20 mg twice daily. In this retrospective study, we compared the efficacy and safety of a quadruple regimen based on low-dose P-CAB (VPZ 20 mg once daily) versus a quadruple regimen based on standard-dose P-CAB (VPZ 20 mg twice daily) or standard-dose proton pump inhibitor (rabeprazole 10 mg twice daily) containing amoxicillin, clarithromycin, and bismuth as initial treatment for H. pylori infection. Our study will provide clinical evidence for the necessary dosage of VPZ in bismuth quadruple regimens, which will help to further optimize the treatment regimen for H. pylori infection.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of H. pylori infection confirmed by urea breath test, monoclonal fecal antigen test, endoscopic biopsy histopathology, or bacterial culture;
2. No previous eradication therapy for H. pylori;
3. Age and gender are not restricted.

Exclusion Criteria:

1. Use of acid-suppressing drugs within 2 weeks prior to treatment, or use of bismuth or antibiotics (including herbal medicines with antimicrobial properties) within 4 weeks prior to treatment;
2. Known hypersensitivity to the drugs used in this study;
3. History of esophageal or gastric surgery;
4. Pregnant or lactating women;
5. Serious systemic diseases, diseases of the heart, lungs, brain and other vital organs, hepatic or renal insufficiency or malignant tumors (except gastric cancer);
6. Patients unable to express their main complaints.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population consisted of patients undergoing initial treatment for H. pylori infection who attended the outpatient clinic of the Department of Gastroenterology at the Second Hospital of Zhejiang University School of Medicine from January 1, 2021 to December 31, 2021. Only patients using a quadruple regimen based on rabeprazole or vonoprazan combined with amoxicillin and clarithromycin with bismuth were included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 558 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Helicobacter H. pylori eradication rate | after eradication therapy at least 4 weeks
  number of patients successfully eradicated / the total number participants

SECONDARY OUTCOMES:
safety of regimens | Within 4 weeks from the beginning to the end of therapy
  comparison of the incidence of adverse events in each group
compliance | 4 weeks after therapy completion
  percentage of correctly administered drugs

CONTACTS AND LOCATIONS:
Overall Officials: Qin DU, Study Chair — Second Affiliated Hospital of Zhejiang University, School of Medicine

IPD SHARING:
Plan to Share IPD: Yes
After the completion of this study, data are available upon reasonable request. Data are available from the corresponding author upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD Sharing will be available from June 30th 2024.
Access Criteria: After the completion of this study, data are available upon reasonable request. Data are available from the corresponding author upon reasonable request.